CLINICAL TRIAL: NCT00480545
Title: Changes in Thrombin Generation Potential and Thromboelastography During the Menstrual Cycle
Brief Title: Changes in Bleeding and Clotting During the Menstrual Cycle
Status: Withdrawn | Type: Observational
Why Stopped: IRB Approval lapsed
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Deborah Brown, Associate Professor - Gulf States Hemophilia Center, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-05-0095
Record Dates: First submitted 2007-05-29; First posted 2007-05-31 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Von Willebrand's Disorder; Healthy
Keywords: Women with bleeding disorders; Menstrual cycle; Women; Healthy volunteers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be discarded when the study is completed.
Oversight: Data Monitoring Committee: No

SUMMARY:
Indirect evidence suggests that hormonal fluctuations during the menstrual cycle also affect the bleeding and clotting system. This study looks at two sensitive laboratory tests at four time points during the menstrual cycle to determine if there is a natural variation in coagulation and platelet function. Laboratory tests in healthy subjects will be compared to women with von Willebrand's disorder type 1, a bleeding disorder. In the future, these laboratory tests may help in the diagnosis of bleeding and clotting disorders and to design treatments for women with abnormal menstrual bleeding.

DETAILED DESCRIPTION:
Von Willebrand disease (VWD) is the most common hereditary bleeding disorder, occurring in 1-2% of the population. Menorrhagia, or heavy menstrual bleeding, occurs in the majority of women with von Willebrand disease (VWD) and adversely affects quality of life. The American College of Obstetrics and Gynecology has recommended that women with heavy menstrual bleeding have diagnostic testing for VWD. Unfortunately, the diagnosis of VWD in women with menorrhagia can be difficult due to fluctuations in hemostatic protein levels during the menstrual cycle. The lack of useful coagulation assays has also limited the scope of pharmacokinetic studies and comparative clinical trials needed to determine best clinical practices in women with VWD.

Two new assay systems offer a possibility of increased sensitivity to physiologic variations in coagulation and fibrinolysis. The calibrated automated thrombin generation assay (TG), an estimation of endogenous thrombin potential (ETP), measures generation of thrombin throughout the entire process of coagulation and has appears to be very sensitive to small changes in levels of coagulation proteins. Thromboelastography (TEG) records clot formation and dissolution in whole blood samples providing a good marker for fibrinolysis. We propose that TG and TEG will be more sensitive than traditional coagulation assays to detect physiologic variations in hemostasis during the menstrual cycle and can accurately diagnose VWD. This is a single-institution pilot study to identify trends which are worthy of further exploration in a larger multi-institutional study. Our primary objective is to describe characteristics of TG and TEG at 4 time points during the menstrual cycle (days 0-3, 7-10, 14-17, and 21-24). Our secondary goal is to quantify the effects of VWD on TG and TEG at the same time points during the menstrual cycle and compare these to traditional coagulation assays.

This will be a single-institution pilot study of a total of 40 subjects: 20 healthy women and 20 women with VWD. Subjects must be female between the ages of 18 and 50 years, have regular menstrual periods, and not be pregnant. Women who are taking hormonal therapy, anti-fibrinolytic therapy, hemostatic agents or anti-platelet agents, will not be eligible for participation. Subjects will be given tampons and/or pads to use during one menstrual cycle. Study participation will involve a brief interview, completion of a questionnaire and a pictorial chart of one menstrual cycle, and having blood drawn at 4 time points during one menstrual cycle. Blood samples will be collected for TG and TEG and standard assays of coagulation and fibrinolysis. TG and TEG measurements will be compared to standard measures of coagulation, fibrinolysis, and platelet activation markers. Serum from the visit on day 21-24 will be tested for progesterone and Bhcg to confirm ovulation and exclude pregnancy. All assays will be performed at the Gulf States Hemophilia & Thrombophilia coagulation laboratory.

This study will result in an improved capability to diagnose women with VWD during the menstrual cycle. These new assays may be useful in the rational design of therapeutic agents and clinical trials. In addition, the physiologic basis of variations in coagulation during the menstrual cycle can be explored in future studies using this assay system.

ELIGIBILITY:
Inclusion Criteria:

* Must be female
* Aged 18 to 50 years, with regular menstrual cycles.
* Healthy volunteers and women with von Willebrand's disorder are both being recruited.

Exclusion Criteria:

* Pregnancy
* Use of hormonal therapy including birth control pills
* Use of hemostatic agents such as DDAVP or anti-platelet agents.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women aged 18 to 50 years with regular menstrual cycles.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Endogenous Thrombin Potential | 28 days
  Changes in coagulation as measured by ETP during the menstrual cycle

SECONDARY OUTCOMES:
von willebrand factor | 28 days
  Changes in von Willebrand factor during the menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L. Brown, M.D., Principal Investigator — University of Texas Health Science Center in Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States